CLINICAL TRIAL: NCT06504121
Title: PFO tRanscatether Occlusion Long-term Outcomes National Group (PROLONG) Registry
Acronym: PROLONG
Status: Completed | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Collaborators: Centro Cardiologico Monzino (Other); University Hospital Padova (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Policlinico Umberto I (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); San Camillo Hospital, Rome (Other); Clinica San Martino (Unknown); University Of Perugia (Other); Maria Cecilia Hospital (Other)
Responsible Party: Principal Investigator, Cosmo Godino, Doctor, IRCCS Ospedale San Raffaele
Other Study IDs: 09031943
Record Dates: First submitted 2024-07-04; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Patent Foramen Ovale; Stroke, Cryptogenic; Transient Ischaemic Attack Due to Embolism; Atrial Fibrillation New Onset
Keywords: Patent Foramen Ovale; Stroke, Cryptogenic; Stroke; Transient Ischemic Attack; Atrial Fibrillation; Interventional cardiology
MeSH Terms: conditions — Foramen Ovale, Patent; Ischemic Stroke; Stroke; Ischemic Attack, Transient; Atrial Fibrillation | interventions — Septal Occluder Device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Device Closure: PFO closure with septal occluder device.
  Interventions: Device: Septal Occluder Device

INTERVENTIONS:
Device: Septal Occluder Device — Transcatheter PFO closure with any commercially available septal occluder device

SUMMARY:
Patent foramen ovale (PFO) has been associated with cryptogenic stroke and transient ischemic attack (TIA) in young adults.

Evidence from randomized clinical trials (RCT) has shown that transcatheter PFO closure yields a 59% relative reduction in recurrent ischemic stroke compared to medical therapy in selected individuals.

However, the follow-up duration in these studies averaged around 4 years, while only two studies report a median follow-up beyond 10 years. Considering the relative youth of the patients undergoing this procedure (average age being under 50 years across all studies), we can reasonably anticipate a substantial post-PFO closure lifespan for these individuals. Consequently, it is imperative to gather more extensive long-term follow-up data among PFO closure recipients The PROLONG (PFO tRanscatether Occlusion Long-term Outcomes National Group) is an observational, retrospective, multicenter, national registry including men and women undergoing transcatheter PFO closure, with the aim of assessing the long-term (>10 years) efficacy and safety of this procedure.

DETAILED DESCRIPTION:
The PROLONG (PFO Transcatheter Occlusion Long-term Outcomes National Group) is an observational, retrospective, multicenter registry. It includes 1,360 subjects who underwent transcatheter patent foramen ovale (PFO) closure between 1999 and 2013 at 12 Italian high-volume Centers. Patients will have at least 10 years of follow-up post-procedure.

The primary objectives of the study are to evaluate the long-term clinical effectiveness of PFO closure by the incidence of left-sided embolic events and to evaluate safety by assessing serious device- or procedure-related adverse events. Secondary objectives include the incidence of new-onset atrial arrhythmias, the presence and severity of residual shunts, the incidence and severity of migraine symptoms, and bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Confirmed Patent Foramen Ovale (PFO);
* Transcatheter Patent Foramen Ovale (PFO) closure with an Occluder device;
* PFO closure procedure performed between 1999 and 2013.

Exclusion Criteria:

* Age < 18 years;
* Previous surgical or transcatheter PFO closure;
* Patients without follow-up data available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The PROLONG registry will enroll a total of 1360 subjects who underwent transcatheter patent foramen ovale (PFO) closure between 1999 and 2013 at 12 high-volume Italian Centers.
  Subjects range in age and gender and encompass individuals from both urban and rural areas, representing a comprehensive sample of patients typically seen in a real-world clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 1360 (Actual)
Dates: Start 1999-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with ischemic stroke, transient ischemic attack or systemic embolism (SE) post device implant (Primary Effectiveness Outcome) | Duration of follow-up (minimum of 10 years)
  The primary effectiveness outcome is the composite incidence of stroke, transient ischemic attack (TIA), and systemic embolism (SE) post-PFO closure.
Number of Participants with device- or procedure-related serious adverse events (Primary Safety Endpoint) | Duration of follow-up (minimum of 10 years)
  Device- or procedure- related serious adverse events post device implant

SECONDARY OUTCOMES:
Number of Participants with recurrent ischemic stroke | Time Frame: Duration of follow-up (minimum of 10 years)
  Incidence of ischemic stroke post-PFO closure.
Number of Participants withrecurrent transient ischemic attack (TIA) | Time Frame: Duration of follow-up (minimum of 10 years)
  Incidence of transient ischemic attack (TIA) post-PFO closure.
Number of Participants with with recurrent systemic embolism (SE) | Time Frame: Duration of follow-up (minimum of 10 years)
  Incidence of systemic embolism (SE) post-PFO closure.
Rate of Procedural Success | Time Frame: Duration of follow-up (minimum of 10 years)
  The rate of successful PFO closure as determined by the absence of severe residual shunt or any procedure- or device-related serious adverse event (SAE)
Incidence of Clinically Significant New Atrial Arrhythmia | Time Frame: Duration of follow-up (minimum of 10 years)
  The occurrence of new-onset atrial fibrillation (AF) or atrial flutter (AFL) following PFO-closure
Rate of All-cause mortality | Time Frame: Duration of follow-up (minimum of 10 years)
  The overall mortality rate of patients post-PFO closure, including both cardiac and non-cardiac causes, documented during follow-up.
Rate of residual shunt | Time Frame: Duration of follow-up (minimum of 10 years)
  Characterization of presence and severity of a residual shunt post-PFO closure, as detected by follow-up echocardiographic assessments.
Incidence of Device-Related and procedure-related Complications | Time Frame: Duration of follow-up (minimum of 10 years)
  The rate of complications related to the PFO closure device, such as device embolization, erosion, or thrombosis, documented during follow-up.
Incidence of bleeding events | Time Frame: Duration of follow-up (minimum of 10 years)
  The rate of bleeding events according to the Bleeding Academic Research Consortium (BARC) criteria
Incidence of migraine symptoms | Time Frame: Duration of follow-up (minimum of 10 years)
  The presence and severity of migraine symptoms will be documented

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pristipino C, Sievert H, D'Ascenzo F, Louis Mas J, Meier B, Scacciatella P, Hildick-Smith D, Gaita F, Toni D, Kyrle P, Thomson J, Derumeaux G, Onorato E, Sibbing D, Germonpre P, Berti S, Chessa M, Bedogni F, Dudek D, Hornung M, Zamorano J; Evidence Synthesis Team; Eapci Scientific Documents and Initiatives Committee; International Experts. European position paper on the management of patients with patent foramen ovale. General approach and left circulation thromboembolism. Eur Heart J. 2019 Oct 7;40(38):3182-3195. doi: 10.1093/eurheartj/ehy649. PMID 30358849
- [Background] Kuijpers T, Spencer FA, Siemieniuk RAC, Vandvik PO, Otto CM, Lytvyn L, Mir H, Jin AY, Manja V, Karthikeyan G, Hoendermis E, Martin J, Carballo S, O'Donnell M, Vartdal T, Baxter C, Patrick-Lake B, Scott J, Agoritsas T, Guyatt G. Patent foramen ovale closure, antiplatelet therapy or anticoagulation therapy alone for management of cryptogenic stroke? A clinical practice guideline. BMJ. 2018 Jul 25;362:k2515. doi: 10.1136/bmj.k2515. No abstract available. PMID 30045912
- [Background] Mendelson SJ, Prabhakaran S. Diagnosis and Management of Transient Ischemic Attack and Acute Ischemic Stroke: A Review. JAMA. 2021 Mar 16;325(11):1088-1098. doi: 10.1001/jama.2020.26867. PMID 33724327
- [Background] Mas JL, Derumeaux G, Guillon B, Massardier E, Hosseini H, Mechtouff L, Arquizan C, Bejot Y, Vuillier F, Detante O, Guidoux C, Canaple S, Vaduva C, Dequatre-Ponchelle N, Sibon I, Garnier P, Ferrier A, Timsit S, Robinet-Borgomano E, Sablot D, Lacour JC, Zuber M, Favrole P, Pinel JF, Apoil M, Reiner P, Lefebvre C, Guerin P, Piot C, Rossi R, Dubois-Rande JL, Eicher JC, Meneveau N, Lusson JR, Bertrand B, Schleich JM, Godart F, Thambo JB, Leborgne L, Michel P, Pierard L, Turc G, Barthelet M, Charles-Nelson A, Weimar C, Moulin T, Juliard JM, Chatellier G; CLOSE Investigators. Patent Foramen Ovale Closure or Anticoagulation vs. Antiplatelets after Stroke. N Engl J Med. 2017 Sep 14;377(11):1011-1021. doi: 10.1056/NEJMoa1705915. PMID 28902593
- [Background] Saver JL, Carroll JD, Thaler DE, Smalling RW, MacDonald LA, Marks DS, Tirschwell DL; RESPECT Investigators. Long-Term Outcomes of Patent Foramen Ovale Closure or Medical Therapy after Stroke. N Engl J Med. 2017 Sep 14;377(11):1022-1032. doi: 10.1056/NEJMoa1610057. PMID 28902590
- [Background] Lee PH, Song JK, Kim JS, Heo R, Lee S, Kim DH, Song JM, Kang DH, Kwon SU, Kang DW, Lee D, Kwon HS, Yun SC, Sun BJ, Park JH, Lee JH, Jeong HS, Song HJ, Kim J, Park SJ. Cryptogenic Stroke and High-Risk Patent Foramen Ovale: The DEFENSE-PFO Trial. J Am Coll Cardiol. 2018 May 22;71(20):2335-2342. doi: 10.1016/j.jacc.2018.02.046. Epub 2018 Mar 12. PMID 29544871
- [Background] Vaduganathan M, Qamar A, Gupta A, Bajaj N, Golwala HB, Pandey A, Bhatt DL. Patent Foramen Ovale Closure for Secondary Prevention of Cryptogenic Stroke: Updated Meta-Analysis of Randomized Clinical Trials. Am J Med. 2018 May;131(5):575-577. doi: 10.1016/j.amjmed.2017.11.027. Epub 2017 Dec 8. PMID 29229471
- [Background] Ahmad Y, Howard JP, Arnold A, Shin MS, Cook C, Petraco R, Demir O, Williams L, Iglesias JF, Sutaria N, Malik I, Davies J, Mayet J, Francis D, Sen S. Patent foramen ovale closure vs. medical therapy for cryptogenic stroke: a meta-analysis of randomized controlled trials. Eur Heart J. 2018 May 7;39(18):1638-1649. doi: 10.1093/eurheartj/ehy121. PMID 29590333
- [Background] Mojadidi MK, Elgendy AY, Elgendy IY, Mahmoud AN, Elbadawi A, Eshtehardi P, Patel NK, Wayangankar S, Tobis JM, Meier B. Transcatheter Patent Foramen Ovale Closure After Cryptogenic Stroke: An Updated Meta-Analysis of Randomized Trials. JACC Cardiovasc Interv. 2017 Nov 13;10(21):2228-2230. doi: 10.1016/j.jcin.2017.09.002. No abstract available. PMID 29122137
- [Background] Wintzer-Wehekind J, Alperi A, Houde C, Cote JM, Asmarats L, Cote M, Rodes-Cabau J. Long-Term Follow-Up After Closure of Patent Foramen Ovale in Patients With Cryptogenic Embolism. J Am Coll Cardiol. 2019 Jan 29;73(3):278-287. doi: 10.1016/j.jacc.2018.10.061. PMID 30678757
- [Derived] Gaspardone C, Trabattoni D, d'Atri DO, Morosato M, Costa P, Fraccaro C, Donti A, Saia F, Toscano E, Scalise F, Cucco A, Patti G, Nerla R, Castriota F, Trani C, Improta R, Mancone M, Sardella G, Musto C, Paciaroni M, Morciano DA, Ricchetti G, Zaccaria L, Beneduce A, Barone G, Salerno A, Vella CS, Montorfano M, Pappone C, Colombo A, Maisano F, Burzotta F, Tarantini G, Margonato A, Gaspardone A, Godino C. 15-Year Outcomes of PFO Closure in Patients With Cryptogenic Embolism: Insights From the PROLONG Registry. JACC Cardiovasc Interv. 2025 Jun 23;18(12):1526-1537. doi: 10.1016/j.jcin.2025.04.041. PMID 40562467